CLINICAL TRIAL: NCT01166659
Title: Study of CyPass Implantation In Patients With Open Angle Glaucoma Refractory to Single or Multi-agent Topical Therapy
Acronym: DUETTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMI-10-03
Record Dates: First submitted 2010-07-14; First posted 2010-07-21 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2016-10

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Glaucoma; Glaucoma device; Glaucoma surgery; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyPass Micro-Stent (Experimental): Subjects receive the CyPass Micro-Stent
  Interventions: Device: CyPass Micro-Stent

INTERVENTIONS:
Device: CyPass Micro-Stent — The CyPass Micro-Stent is a small tube with a through-lumen designed to redirect aqueous fluid from the front to the back of the eye. The CyPass is implanted in the eye.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CyPass implantation as a stand-alone therapy for lowering intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) who have failed at least one class of topical medical therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG
* Medicated IOP ≥ 21 and ≤ 35 mmHg
* Use of 1 - 4 topical IOP lowering medications

Exclusion Criteria:

* Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma
* Use of oral hypotensive medication treatment for glaucoma
* Previous incisional glaucoma surgery, or any combined cataract-glaucoma procedure
* Clinically significant ocular pathology other than POAG

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President of Medical Affairs, Study Chair — Transcend Medical, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 investigational sites in Germany, Bulgaria, Spain and Austria.
Pre-assignment Details: This reporting group includes all treated participants.
Groups:
- CyPass Micro-Stent: Subjects received the CyPass Micro-Stent
Period: Overall Study
Arm/Group | CyPass Micro-Stent
Started | 48
Completed | 35
Not Completed | 13
Not completed — Subject Decision | 8
Not completed — Investigator Decision | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Study Closed at Site | 1

BASELINE CHARACTERISTICS:
Arm/Group | CyPass Micro-Stent
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 16
Region of Enrollment [Number; unit: participants]
  Austria | 4
  Bulgaria | 8
  Germany | 33
  Spain | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Intraocular Pressure (IOP) Reduction of ≥ 20% at 12 Months Postoperatively Who Were on Fewer or the Same Number of Ocular Hypotensive Medications as Compared With Baseline
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). A reduction in IOP from baseline indicates an improvement. Proportion of eyes is reported as a percentage.
Time Frame: Baseline; Month 12 postoperative
Population: Eyes implanted with the CyPass 2FX device with data available.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass Micro-Stent
Number analyzed (Participants) | 42
Number analyzed (eyes) | 43
percentage of eyes | 60.4

2. Secondary Outcome: Proportion of Eyes With Achievement of Target IOP With and Without Use of Ocular Hypotensive Medication
Description: Target IOP was defined as ≥ 6 mmHg and ≤ 21 mmHg. Proportion of eyes is reported as a percentage.
Time Frame: Month 12 postoperative
Population: Eyes implanted with the CyPass 2FX device with data available.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass Micro-Stent
Number analyzed (Participants) | 42
Number analyzed (eyes) | 43
percentage of eyes | 81.4

3. Secondary Outcome: Mean Number of Topical IOP-Lowering Medications Used in Comparison With Baseline
Description: The number of unique glaucoma medications was recorded. The mean number of topical IOP-lowering medications was computed by dividing the total number of medications used (the numerator) by the total number of subjects who reported on medication use at the visit.
Time Frame: Baseline, Month 12 postoperative
Population: Eyes implanted with the CyPass 2FX device with data available.
Measure: Mean (Standard Deviation); unit: medications
Units Other Than Participants: eyes
Arm/Group | CyPass Micro-Stent
Number analyzed (Participants) | 42
Number analyzed (eyes) | 43
medications
  Baseline | 2.1 (0.99)
  Month 12 | 1.4 (1.3)

ADVERSE EVENTS:
Time Frame: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury or any untoward clinical sign occurring in a study subject, whether or not related to the CyPass device. AEs were collected from time of consent to study exit (Month 24 postoperative).
Description: Reports of AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Non-Ocular Adverse Events: At risk population for non-ocular adverse events is included with unit of subjects
- Ocular Adverse Events: At risk population for ocular adverse events is included with unit of eyes.
Arm/Group | Non-Ocular Adverse Events | Ocular Adverse Events
Serious Adverse Events (participants affected / at risk) | 2/48 | 8/50
Other Adverse Events (participants affected / at risk) | 0/48 | 36/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Ocular Adverse Events (N=48) | Ocular Adverse Events (N=50)
Secondary surgical intervention (Injury, poisoning and procedural complications) | 0 | 3
IOP above target (Investigations) | 0 | 5
Death (General disorders) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Ocular Adverse Events (N=48) | Ocular Adverse Events (N=50)
Hyphema (Eye disorders) | 0 | 3
BCVA loss ≥ 2 lines at/after 3 months postoperatively (Eye disorders) | 0 | 12
Secondary surgical intervention: IOP management (Injury, poisoning and procedural complications) | 0 | 13
IOP ≥ 10 mmHg over baseline or > 30 mmHg at/after 1 month postoperatively (Investigations) | 0 | 10
CyPass device obstruction (Investigations) | 0 | 6
Secondary surgical intervention: Cataract removal (Injury, poisoning and procedural complications) | 0 | 11
Secondary surgical intervention: CyPass obstruction lysis (Injury, poisoning and procedural complications) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.